CLINICAL TRIAL: NCT06708130
Title: Allogeneic Hematopoietic Stem Cell Transplantation Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Xiaoxia, Director of the Center for Translational Medicine, Ruijin Hospital
Other Study IDs: RJ-BMT
Record Dates: First submitted 2024-11-13; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Patients who are proposed to undergo or have undergone allogeneic hematopoietic stem cell transplantation at the Stem Cell Transplant Center and Post-Transplant Medical Consortium at Regent Hospital

SUMMARY:
Clinical observational studies using epidemiologic theories and methods. Through the collection of various clinically relevant data, specific outcomes are evaluated in hematologic transplant patients, providing high quality real-world data for clinical practice, informing public health decision-making, and reducing the burden of disease

DETAILED DESCRIPTION:
This is a retrospective, prospective, two-way cohort study in which clinical diagnostic and treatment data will be collected on patients enrolled in the study and followed up to characterize the natural course of the patient population as systematically as possible. All treatment decisions and clinical assessments will be made by the treating physician based on conventional treatment criteria and are not required by the study design or protocol.

The purpose of this study is to examine the natural course of the disease and current treatments. An in-depth analysis of treatment regimens and treatment duration, as well as the sequence of regimen use, will be conducted to describe treatment modalities and healthcare expenditures for this disease state. No clinical device or laboratory/assessment interventions will be conducted except for disease management requirements based on routine practice requirements or treatment monitoring based on locally approved product characterization requirements. Patients will be required to complete a separate questionnaire containing basic epidemiologic information (demographics, disease history, environmental exposure history).

During the duration of this study, some patients may be enrolled in interventional clinical trials. This is allowed and expected to occur in this study. Patients will not be required to withdraw from the cohort study and will continue to be followed up as normal, unless the investigator/patient feels it is more appropriate to withdraw from the study. All requirements of the clinical trial in question are documented according to the trial protocol.

ELIGIBILITY:
Inclusion Criteria:

1. At least one visit to a stem cell transplant center beginning January 1, 2021
2. Proposed to undergo or have undergone hematopoietic stem cell transplantation

Exclusion Criteria:

1. Long-term follow-up information for patients not available for any reason (e.g., unavailable or with serious concomitant disease) according to investigator opinion
2. Due to alcohol and drug addiction thus affecting their ability to follow the requirements of the study
3. Presence of conditions that could jeopardize patient safety or affect their adherence to the protocol, according to the investigator's opinion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are proposed to undergo or have undergone allogeneic hematopoietic stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Time Frame: through study completion, an average of 5 year
  OS since enrollment

SECONDARY OUTCOMES:
Strictly complete remission (sCR) | Time Frame: through study completion, an average of 5 year
  Strictly complete remission (sCR)
Complete remission (CR) | Time Frame: through study completion, an average of 5 year
  Complete remission (CR)
Very Good Partial Relief (VGPR) | Time Frame: through study completion, an average of 5 year
  Very Good Partial Relief (VGPR)
Partial remission (PR) | Time Frame: through study completion, an average of 5 year
  Partial remission (PR)
Minor Relief (MR) | Time Frame: through study completion, an average of 5 year
  Minor Relief (MR)
Disease stabilization (SD) | Time Frame: through study completion, an average of 5 year
  Disease stabilization (SD)
Progression of Disease (PD) | Time Frame: through study completion, an average of 5 year
  Progression of Disease (PD)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Liquan Hospital, Shanghai
  - Shanghai Zhaxin Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No